CLINICAL TRIAL: NCT02385747
Title: Assessment of Uterine Cavity and Endometrial Steroid Receptors in Women With Peri- and Post Menopausal Bleeding
Brief Title: Uterine Cavity Assessment and Endometrial Hormonal Receptors in Women With Peri and Post Menopausal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 130
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Vaginal Bleeding
Keywords: perimenopausal bleeding; postmenopausal bleeding; hysteroscopy; Steroid receptors
MeSH Terms: conditions — Uterine Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- women with anbormal bleeding (Experimental): women with perimenopausal and postmenopausal bleeding who will be evaluated with transvaginal ultrasound, saline sonohysterography,hystroscopy and endometrial currettage
  Interventions: Procedure: hystroscopy

INTERVENTIONS:
Procedure: hystroscopy — Detailed hysteroscopic examination under general anesthesia Once the cavity entered, a panoramic view of the uterine cavity then systematic; first the fundus, then anterior, posterior and lateral walls of the uterus consecutively, ending by visualization of the uterine -tubal junctions, The thickness, colour, aspect and vasculature of the mucous membrane lining the uterine cavity was observed and recorded. If there is any intrauterine pathology detected; the shape, size and site were estimated.

SUMMARY:
100 women with abnormal uterine bleeding (peri and postmenopausal) were subjected to transvaginal ultrasound , saline sonohysterography , Diagnostic hysteroscopy and fractional curettage followed by histopathological examination and immunohistochemical analysis for estrogen and progesterone receptors.

DETAILED DESCRIPTION:
Conventional TVUS will be done to all participants to measure the uterine size & endometrial thickness and other pathology. TVUS will be done with an empty bladder in the lithotomy position using an endovaginal curved linear probe (EV 4-9/10 ED) with frequency 4-9 MHz.

SIS will be performed for all patients at the same setting of TVUS. With the patient in the lithotomy position, . A 6 or 8 French Foley's catheter will be inserted through the external cervical os into the cervical canal. Its balloon tip will be inflated with 2-3 mL of saline, depending on patient comfort, to help hold it in place. The speculum was then removed.

The vaginal probe was then reinserted and a 5-10 mL syringe filled with sterile saline was attached to the catheter. Fluid will be instilled while the transducer moved from side to side (cornua to cornua) in a long-axis projection then the transducer was rotated 90° into an axial plane. More fluid was instilled while fanning down toward the endocervical canal and up toward the uterine fundus to obtain a detailed survey of the endometrium. Every portion of the uterine cavity should be imaged, to exclude any focal abnormality as polyps, myomas, hyperplasia, and carcinoma. Any detected intrauterine pathology is described; including its shape, size and site.

The hysteroscope used in this study is a rigid continuous flow panoramic hysteroscope, 25 cm in length, 4 mm in diameter with an outer sheath 5 mm diameter and 30° fibro-optic lens.

The technique used to provide constant uterine distention will be by attaching plastic bags of saline. Infusion pressure was elevated by pneumatic cuff under manometric control at a pressure of 100-120 mmHg.

Detailed hysteroscopic examination will be performed under general anesthesia with the patient in the lithotomy position, The thickness, colour, aspect and vasculature of the mucous membrane lining the uterine cavity will be observed and recorded.

Endometrial curettage will be done to all patients, and specimens were fixed in Formalin 10% solution for histopathological examination. Patients in whom endometrial polyps were found by hysteroscopy, had polypectomy performed before curettage. The first sample will be taken from the endocervical canal before hysteroscopy or cervical dilatation. Following diagnostic hysteroscopy, cervical dilatation u. A sharp curette will be introduced into the uterine cavity, and curettage will be done starting with the fundus then posterior, anterior, right and left lateral walls consecutively.

Histopathological examination. All curettage & polypectomy specimens were embedded in paraffin wax, then slides will be prepared to be stained by the conventional Haematoxylin and Eosin (H & E) stain.

Detection of estrogen & progesterone receptors in the specimens (formalin-fixed, paraffin wax-embedded) using immunohistochemical staining which will be carried out by using the Dako ER/PR pharmDx™ Kit which specifically detects the ERα protein as well as the PR-A protein located in the cell nuclei of ER and PR expressing cells, respectively.

ELIGIBILITY:
Inclusion Criteria:

* women older than 45 years with Abnormal uterine bleeding for more than 3 months duration

Exclusion Criteria:

* history of hormonal treatment or hormonal contraception within the last 6 months. Women who had used IUD or those had hysteroscopy or fractional curettage done within the last 6 months

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
detection of endometrial lesion | 2 days after curretage

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt